CLINICAL TRIAL: NCT04107649
Title: Knee Arthroplasty Activity Trial
Acronym: KArAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Northwestern Memorial Hospital (Other); University of Kansas Medical Center (Other); University at Buffalo (Other); University of Nebraska (Other)
Responsible Party: Principal Investigator, Elena Losina, Co-Director of OrACORe, Robert W. Lovett Professor of Orthopaedic Surgery at Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019P002700
Record Dates: First submitted 2019-09-24; First posted 2019-09-27 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis; Total Knee Replacement
Keywords: Physical Activity; Total Knee Replacement; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Three arm parallel randomized control trial.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigators, care providers, and outcomes assessors will not be appraised of treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm1 (Other): Participants in this arm receive usual post-operative care and complete all basic study activities, which include: attending 2 in-clinic visits at designated time-points, having regular check-in calls with study staff over the intervention period, wearing and returning waist-worn activity trackers at 5 time points over two years, and completing 6 study surveys.
  Interventions: Other: Basic Study Activities
- Arm2 (Experimental): Participants in this arm receive usual post-operative care, complete all basic study activities (as described in arm 1) and receive the wrist-based activity tracker intervention.
  Interventions: Behavioral: Wrist based activity tracker wear; Other: Basic Study Activities
- Arm3 (Experimental): Participants in this arm receive usual post-operative care, complete all basic study activities (as described in arm 1), receive wrist-based activity tracker intervention, and receive the TAC(MI)+FI.
  Interventions: Behavioral: Telephonic Active Coaching (Motivational Interviewing) + Financial Incentives; Behavioral: Wrist based activity tracker wear; Other: Basic Study Activities

INTERVENTIONS:
Behavioral: Telephonic Active Coaching (Motivational Interviewing) + Financial Incentives — As part of TAC(MI)+FI, participants speak with a health coach at Brigham and Women's Hospital once a week via telephone for weeks 6-13 following surgery, and once every other week for weeks 14-31 after surgery. Participants in this arm can receive financial rewards for achieving weekly physical activity goals, as well as bonus rewards for achieving goals multiple weeks in a row. Over the course of this 6-month long TAC(MI)+FI intervention period, these participants are able to receive up to $680 for meeting physical activity goals, and up to $95 in bonus rewards.
  Other Names: TAC(MI)+FI
  Arms: Arm3
Behavioral: Wrist based activity tracker wear — Activity tracking data will be collected on a weekly basis. Participants who receive this intervention are eligible to be entered into a lottery to win one of two $25 rewards for every week they wear their wrist-based activity tracker >10 hours for >4/7 days a week, beginning 6-weeks after surgery.
  Arms: Arm2; Arm3
Other: Basic Study Activities — Basic study activities begin two-weeks before TKR and end approximately 24-months after TKR. Basic study activities include: two in-person visits at the local clinic site (2 weeks before TKR and 32-weeks after TKR), having check-in calls with study staff weekly from weeks 1-13 after surgery and every other week for weeks 14-31, completing 6 surveys, and wearing an ActiGraph activity tracker (waist-worn) for five one-week periods throughout the study (2-weeks before-TKR, 32-weeks post-TKR, one-year post-TKR, 18-months post-TKR, two-years post-TKR). All participants will be eligible to receive up to $235 for completing these activities over the course of two years.

SUMMARY:
Total knee replacement (TKR) is a common and costly procedure widely used to relieve pain and improve function in patients with symptomatic advanced knee osteoarthritis (OA). As of 2013, the annual incidence of TKR was over 680,000 surgeries and annual costs exceeded $11 billion. Growing evidence suggests that while pain and functional status improve following TKR, physical activity (PA) typically does not surpass pre-TKR levels. Engagement in PA can meaningfully improve quality of life (QoL), pain, and function. Given the large investment in TKR, the effectiveness and cost-effectiveness of TKR could be substantially increased if TKR recipients became more physically active.

The Knee Arthroplasty Activity Trial (KArAT) is a randomized controlled trial and participants will be randomly assigned to one of three arms. Participants across all arms will receive usual post-operative care for TKR surgery. Participants in the first arm will complete basic study activities, such as responding to surveys and attending two in-person clinic visits. Participants in the second arm will do the same and also receive a wrist-based physical activity tracker intervention. Participants in the third arm will receive a telephonic active coaching (motivational interviewing) and financial incentives (for reaching physical activity goals) (TAC(MI)+FI) based intervention, as well as a wrist-based physical activity tracker intervention. The second and third arms will be eligible to receive lottery-based financial rewards for wearing a wrist-worn activity tracker for twenty-four months during the study.

DETAILED DESCRIPTION:
The investigators have designed the KArAT trial with two specific aims. First, to conduct a parallel three-arm RCT to establish the efficacy and sustainability of the effect of personalized intervention built on the principles of behavioral science and behavioral economics in improving PA among sedentary people who have undergone TKR. Our second aim is to establish the cost-effectiveness and budget impact of TAC(MI)+FI to improve PA in persons who have undergone TKR.

The three arms will include:

Arm 1: Usual post-TKR care

Arm 2: Usual post-TKR care + Wrist-based physical activity tracker wear

Arm 3: Usual post-TKR care + Wrist-based physical activity tracker wear + Telephonic Active Coaching (Motivational Interviewing) + Financial Incentives (TAC(MI)+FI).

ELIGIBILITY:
Inclusion Criteria:

* Age 40-85 years
* English-speaking
* Scheduled to undergo primary, unilateral total knee replacement (TKR) at one of the 4 recruitment centers
* OA is principal underlying indication for TKR
* During an accelerometer run-in period lasting one week at baseline (prior to surgery), subjects must show that they can comply with waist-worn physical activity tracker protocols by wearing the activity tracker for ≥4/7 days of the week for ≥10 hours/day
* Regular access to a personal computer, laptop, tablet, or smartphone for wrist-worn activity tracker syncing
* Satisfying average baseline steps/day criteria (calculated from waist-worn activity tracker data from the run-in period)

Exclusion Criteria:

* Non-English speaking
* Residence in nursing home
* Diagnosis of dementia, epilepsy, Parkinson's Disease, or diabetes with peripheral neuropathy
* Inflammatory arthritis (rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, reactive arthritis, systemic lupus erythematosus, polymyalgia)
* Psychological issues that preclude participation
* Inpatient or other musculoskeletal surgery scheduled within six months following index primary TKR
* Uses a wheelchair to ambulate (subjects who use a cane will be eligible)
* Surgeon-documented other reason for study exclusion
* Subject does not have regular access to a device capable of receiving email or text messages

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2028-06-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of Subjects Engaged in at least 150 min/week of moderate-to-vigorous physical activity (MVPA). | 32-weeks post-TKR
  The primary outcome of this trial is the proportion of subjects who meet or surpass the PA threshold of 150 minutes per week of at least moderate physical activity, which is defined as 3 metabolic equivalents (METs), at 32-weeks post-TKR.

SECONDARY OUTCOMES:
Change in average daily step count | 2-week pre-TKR to 32-weeks post-TKR
  Change in subjects' average daily step count from pre-TKR to 32-weeks post-TKR as measured by the ActiGraph.
Change in weekly minutes of moderate-to-vigorous activity (MVPA) | 2 week pre-TKR to 32-weeks post-TKR
  Change in the number of minutes per week that subjects spend engaged in MVPA from pre-TKR to 32-weeks post-TKR as measured by the ActiGraph.
Change in average daily sedentary time | 2 weeks pre-TKR to 32-weeks post-TKR
  Change in subjects' daily sedentary time from pre-TKR to 32-weeks post-TKR as measured by the ActiGraph.

OTHER OUTCOMES:
Durability of changes in activity levels | 2 weeks pre-TKR to 24 months post-TKR
  Changes in subjects' activity levels at 12-, 18-, and 24-months post-TKR as measured by the ActiGraph.
Change in pain and functional status | 2 weeks pre-TKR to 24 months post-TKR
  Change in subjects' pain and functional status at 8-, 12-, 18-, and 24-months post-TKR as measured by the questionnaire.
Change in quality of life | 2 weeks pre-TKR to 24 months post-TKR
  Change in subjects' quality of life at 8-, 12-, 18-, and 24-months post-TKR as measured by the questionnaire.
Change in performance measures | 2 weeks pre-TKR to 6 months post-TKR
  Change in subjects' performance at 32 weeks post-TKR as measured by performance tests.
Change in cost | 2 weeks pre-TKR to 24 months post-TKR
  Change in subjects' medical costs at 8-, 12-, 18-, and 24-months post-TKR as measured by the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Losina, Ph.D., Principal Investigator — Brigham and Women's Hospital
Locations (5):
- United States (5):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University at Buffalo, Buffalo, New York

REFERENCES:
- [Derived] Losina E, Collins JE, Kumara M, Ehrlich-Jones L, Opare-Addo M, Safran-Norton C, Segal NA, Mitchell LM, Kopp PT, Selzer F, Mass H, Paskewicz M, Chang RW, Dunlop D, Chen AF, Lerner S, Chin S, Pellegrini C, Katz JN. KArAT (Knee Arthroplasty Activity Trial): Rationale and design features of a multicenter randomized controlled trial. Osteoarthr Cartil Open. 2024 Aug 23;7(2):100512. doi: 10.1016/j.ocarto.2024.100512. eCollection 2025 Jun. PMID 40276263